CLINICAL TRIAL: NCT00217152
Title: An Open Label, Prospective, Randomized, Controlled, Multicenter Study Assessing Fixed Dose vs. Concentration Controlled CellCept Regimens for Patients Following a Single Organ Renal Transplantation in Combination With Full Dose and Reduced Dose Calcineurin Inhibitors
Brief Title: A Kidney Transplant Study to Look at the Effects of Taking Fixed Doses of CellCept Versus Taking Doses of CellCept Based on the Concentration of CellCept in the Blood When Taking Full or Reduced Dose Calcineurin Inhibitors
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Roche decided to prematurely terminate study.
Sponsor: Mayo Clinic (Other)
Collaborators: Roche Pharma AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112-05
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Kidney Transplantation; Delayed Graft Function
Keywords: Kidney Transplant
MeSH Terms: conditions — Delayed Graft Function | interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: CellCept

SUMMARY:
This research is being done to study the effects (good and bad) of taking CellCept based on blood concentrations versus taking a fixed dose of CellCept without measuring the blood concentration. CellCept is one of the three immunosuppressant drugs (drugs that suppress the immune system) which will be taken as part of this kidney transplant study. Cyclosporine or tacrolimus and corticosteroids are the two other drugs which will be taken.

DETAILED DESCRIPTION:
This study is an open label study, which means the participant will know which drugs they are on. Participants will be put in one of three groups within 24 hours of the participant's transplant. The participant will be asked to return throughout the 24 months for physical exams, blood and urine tests.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 18 and 70 years of age and should be receiving their first or second kidney transplant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-03; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Treatment failure defined as a biopsy proven acute rejection, graft loss, death, or lost to follow-up | during the first 12 months following randomization
Assessment of renal function | 12 months post randomization

SECONDARY OUTCOMES:
The proportion of patients experiencing biopsy proven acute rejections
The total number of biopsy proven, acute rejection episodes, per patient
The proportion of patients treated for acute rejection
The time to the first proven acute rejection
The time to the treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Stegall, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States